CLINICAL TRIAL: NCT05212038
Title: An Iliopsoas Plane Block for Pain Management After Total Hip Arthroplasty: a Randomized Controlled Trial
Brief Title: An Iliopsoas Plane Block After Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Do-Hyeong Kim, Associate Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 3-2021-0438
Record Dates: First submitted 2022-01-11; First posted 2022-01-27 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Total Hip Arthroplasty

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- liopsoas plane block group (Experimental): Arm Description: a iliopsoas plane block before surgery
  Interventions: Procedure: iliopsoas plane block group
- sham block group (Sham Comparator): sham block before surgery
  Interventions: Procedure: sham block group

INTERVENTIONS:
Procedure: iliopsoas plane block group — Ultrasound-guided iliopsoas plane block with 0.75% ropivacaine 10 ml and epinephrine 0.05 ml (1:200,000) 10 ml
  Arms: liopsoas plane block group
Procedure: sham block group — Ultrasound-guided iliopsoas plane block with normal saline 10 ml
  Arms: sham block group

SUMMARY:
Nielsen et al. reported that when iliopsoas plane block was performed on healthy volunteers, the injection solution in Hip MRI was confined to the myofascial compartment, which was known to include all sensory branches of the femoral nerve that control the hip joint. The maximal muscle strength of knee extension did not decrease before and after Iliopsoas plane block in Volunteer. Since there is no clinical study conducted on patients after the volunteer study, the investigators intend to evaluate the analgesic and motor preserving effects of the iliopsoas plane block in a group of patients undergoing total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 19 years of age or older who are expected to undergo unilateral hip arthroplasty
2. ASA PS 1-3

Exclusion Criteria:

1. Revision total hip arthroplasty
2. Allergy to drugs used in the study
3. Patients with moderate or more hepatic impairment (AST/ALT is more than 2.5 times the upper limit of normal)
4. Estimated glomerular filtration rate < 30 mL/min/1.73m2
5. Opioid dependence
6. Prolongation of PT and aPTT more than twice the upper limit of normal
7. Pre-existing neurological or anatomical disorders of the lower extremities
8. Serious psychiatric disorders

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale pain score at rest | up to 48 hours after the surgery
  Pain intensity at rest will be evaluated by an 11-point numeric rating scale (NRS: 0 = no pain, 10 = worst imaginable pain) 1, 6, 24, and 48 hours after the surgery.

SECONDARY OUTCOMES:
Numeric rating scale pain score at movement | up to 48 hours postoperatively
  Pain intensity during 45-degree passive flexion of the hip with the ipsilateral knee flexed naturally will be evaluated by an 11-point numeric rating scale (NRS: 0 = no pain, 10 = worst imaginable pain) 1, 6, 24, and 48 hours after the surgery.
Postoperative opioid consumption | postoperative 24, 48hours
  morphine equivalent dose

CONTACTS AND LOCATIONS:
Locations (1):
- Ji Yeong Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim JY, Lee JS, Kim JY, Yoon EJ, Lee W, Lee S, Kim DH. Iliopsoas plane block does not improve pain after primary total hip arthroplasty in the presence of multimodal analgesia: a single institution randomized controlled trial. Reg Anesth Pain Med. 2025 Mar 5;50(3):257-263. doi: 10.1136/rapm-2023-105092. PMID 38286736